CLINICAL TRIAL: NCT02453841
Title: Prospective Hemodynamic and Pharmacokinetic Analysis of Oxymetazoline Absorption During Functional Endoscopic or Turbinate Reduction Surgery or Adenoidectomy
Brief Title: Prospective Hemodynamic and Pharmacokinetic Analysis of Oxymetazoline Absorption
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Richard Cartabuke (Other)
Responsible Party: Sponsor-Investigator, Richard Cartabuke, Co-Director of Outpatient Anesthesia Services, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB14-00723
Record Dates: First submitted 2015-05-15; First posted 2015-05-27 (Estimated); Results first posted 2018-09-18 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Adenoidectomy; Functional Endoscopic Sinus Surgery (FESS); Turbinate Surgery
MeSH Terms: interventions — Oxymetazoline

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- FESS (Active Comparator): Patients undergoing functional endoscopic sinus surgery and receiving oxymetazoline as part of their surgery.
  Interventions: Drug: Oxymetazoline
- Turbinates (Active Comparator): Patients undergoing turbinate reduction surgery and receiving oxymetazoline as part of their surgery.
  Interventions: Drug: Oxymetazoline
- Adenoidectomy (Active Comparator): Patients undergoing an adenoidectomy and receiving oxymetazoline as part of their surgery.
  Interventions: Drug: Oxymetazoline

INTERVENTIONS:
Drug: Oxymetazoline
  Other Names: Afrin

SUMMARY:
This proposed study will assess the hemodynamic effects and measure the systemic absorption of topically applied oxymetazoline in patients undergoing functional endoscopic sinus surgery, turbinate surgery, or adenoidectomy. These patients will be receiving oxymetazoline as standard of care during the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients that are scheduled for:

  1. Functional endoscopic sinus surgery
  2. Turbinate reduction (with or without tonsillectomy and/or adenoidectomy)
  3. Adenoidectomy

Exclusion Criteria:

* Been treated with oral decongestants or antihistamines within 24 hours of surgery
* Are taking anticoagulants
* Have a history of nasal trauma
* Have a history of epistaxis
* Have a history of hypertension or cardiac disease
* Allergy to oxymetazoline

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2015-12; Primary Completion 2017-04-20 (Actual); Study Completion 2017-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Cartabuke, MD, Principal Investigator — Nationwide Children's Hospital
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Children Undergoing ENT Surgery: Pediatric patients undergoing functional endoscopic sinus surgery (FESS), turbinate surgery, adenoidectomy or a combination of any of these.
Period: Overall Study
Arm/Group | Children Undergoing ENT Surgery
Started | 30
Completed | 27
Not Completed | 3
Not completed — Protocol Violation | 1
Not completed — Unable to obtain blood samples | 2

BASELINE CHARACTERISTICS:
Arm/Group | Children Undergoing ENT Surgery
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 30
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7 (4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 22
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Following Oxymetazoline Administration
Description: Blood pressure was recorded at 5 minute intervals until discharge from the post-anesthesia care unit (PACU) or the final blood draw (150 mins. after administration), whichever came first.
Time Frame: 5 - 150 mins. after administration
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Children Undergoing ENT Surgery
Number analyzed (Participants) | 27
mmHg
  Systolic blood pressure | 102 (16)
  Diastolic blood pressure | 53 (17)
  Mean arterial pressure | 65 (15)

2. Primary Outcome: Heart Rate Following Oxymetazoline Administration.
Description: Heart rate was recorded at 5 minute intervals until discharge from the post-anesthesia care unit (PACU) or the final blood draw (150 mins. after administration), whichever came first.
Time Frame: 5 - 150 mins. after administration
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Children Undergoing ENT Surgery
Number analyzed (Participants) | 27
beats per minute | 98 (22)

3. Secondary Outcome: Ease of Hemostasis
Description: A six point scale (very easy, easy, usual, some effort, difficult, extremely difficult) completed by the surgeon at the end of surgery.
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Children Undergoing ENT Surgery
Number analyzed (Participants) | 27
Participants
  Very Easy | 10
  Easy | 9
  Usual | 8

4. Secondary Outcome: Amount of Bleeding
Description: A four point scale (none, minimal, moderate/diffuse ooze, severe/brisk) completed by the surgeon after removal of the oxymetazoline soaked pledgets.
Time Frame: intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | Children Undergoing ENT Surgery
Number analyzed (Participants) | 27
Participants
  None | 11
  Minimal | 11
  Moderate | 5

ADVERSE EVENTS:
Time Frame: Until discharge from hospital, approximately 24 hours.
Arm/Group | Children Undergoing ENT Surgery
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-03-05): https://cdn.clinicaltrials.gov/large-docs/41/NCT02453841/Prot_SAP_ICF_000.pdf